CLINICAL TRIAL: NCT00214045
Title: Rigid Versus Flexible Cystoscopy in Women in Outpatient Clinic
Brief Title: Rigid Versus Flexible Cystoscopy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-2004-0254; NCT00590733 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Hematuria; Urination Disorders; Voiding Dysfunction; Recurrent Urinary Tract Infection
Keywords: Bladder cancer surveillance; Voiding dysfunction; Cystoscopy
MeSH Terms: conditions — Hematuria; Urination Disorders; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible Cystoscopy (Active Comparator): Flexible Cystoscopy
  Interventions: Device: Flexible Cystoscopy
- Rigid Cystoscopy (Active Comparator): Rigid Cystoscopy
  Interventions: Device: Rigid Cystoscopy

INTERVENTIONS:
Device: Flexible Cystoscopy
  Arms: Flexible Cystoscopy
Device: Rigid Cystoscopy
  Arms: Rigid Cystoscopy

SUMMARY:
The study will help define the best tolerated approach to cystoscopy in women by randomly comparing flexible to rigid cystoscopy. Previous randomized studies evaluated rigid cystoscopy under general anesthesia versus flexible cystoscopy under local anesthesia. As a result of these studies, flexible cystoscopy is performed in the clinic setting generally in males. However, many women have rigid cystoscopy performed in the clinic while the men have flexible cystoscopy. No studies to date have evaluated whether flexible cystoscopy is better tolerated in women compared to rigid cystoscopy in women in the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Female

Exclusion Criteria:

* Minors
* Incarcerated individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nakada, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flexible Cystoscopy: Use of Flexible Cystoscope during clinically indicated cystoscopy
- Rigid Cystoscopy: Use of Rigid Cystoscope during clinically indicated cystoscopy
Period: Overall Study
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Number; unit: participants]
  Minors, <18 yrs | 0 | 0 | 0
  Adults, >=18 yrs | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale for Pain
Description: The Visual Analog Scale for pain ranges from 1 to 5, with higher scores indicating higher pain. Results report the average of two measures, taken during procedure and 1 week post-procedure.
Time Frame: During procedure and 1 week post-procedure
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Rigid: Rigid
- Flexible: Flexible
Arm/Group | Rigid | Flexible
Number analyzed (Participants) | 18 | 18
Units on a Scale | 1.8 (0.2) | 1.4 (0.3)
Statistical Analysis 1: Comparison: Rigid vs Flexible; Test type: Superiority or Other — Results were analyzed using Wilcoxon rank sums and Fisher exact tests with Statistical Analysis System (SAS) statistical software version 9; p = .39, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rigid vs Flexible; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.37, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Flexible Cystoscopy | Rigid Cystoscopy
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes